CLINICAL TRIAL: NCT04462172
Title: A Prospective Multicenter Cohort Study About Internal Fixation Using Synthes Femoral Neck System (FNS) Versus Multiple Cancellous Screws (MCS) for Femoral Neck Fracture
Brief Title: A Prospective Multicenter Cohort Study About Internal Fixation Using FNS Versus MCS for Femoral Neck Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Beijing Jishuitan Hospital (Other); Shanghai 6th People's Hospital (Other); Tianjin Hospital (Other); The Fuzhou No 2 Hospital (Other); Xi'an Honghui Hospital (Other); West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUTH ZF FNS
Record Dates: First submitted 2020-06-28; First posted 2020-07-08 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-06

CONDITIONS: Femoral Neck Fractures
Keywords: femoral neck fracture; internal fixation; FNS and MCS; multicenter randomized controlled clinical trial; internal fixation failure rate
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Intervention Model Description: This prospective multicenter cohort study is to compare the post-operative implant failure rate between the patients with femoral neck fracture (AO classification 31-B) using Femoral Neck System (FNS) versus Multiple Cancellous Screws (MCS) at 2-year follow up.The patients are divided into the FNS group and the MCS group according to the internal fixation they choose.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Synthes Femoral Neck System (FNS) (Experimental): Synthes Femoral Neck System (FNS) was developed with the intention to combine advantages of DHS (dynamic hip screw) and MCS (multiple cancellous screw). The FNS implants consist of plates, bolts, locking screws and antirotating-screws. The plate consists of a small base plate with one or two locking holes and a barrel portion. The barrel allows for gliding of the head elements while restricting rotation around the head-neck axis, so FNS is a fixed-angle gliding fixation device that allows for controlled collapse of the femoral neck, like DHS. The FNS was also designed to minimize implant footprint on the bone with its compact design, like MCS. Furthermore, the FNS was designed to reduce the length of incision necessary for implant insertion when compared to DHS. This new concept of femoral neck fracture fixation still emphasizes the biology of fracture healing by initial fracture compression.
  Interventions: Device: FNS
- Multiple cancellous screws (MCS) (Active Comparator): Multiple cancellous screws (MCS) fixation is the most common and classic method to deal with femoral neck fractures which is less invasive and retains more viable bone, compared with dynamic hip screw (DHS) fixation that appears biomechanically more stable. In this study, three cancellous screws with an inverted triangle pattern are used to fix the fracture of femoral neck.
  Interventions: Device: MCS

INTERVENTIONS:
Device: FNS — perform preoperative preparation, intraoperative operation and internal fixation implantation according to the instructions provided in the product packaging.
  Arms: Synthes Femoral Neck System (FNS)
Device: MCS — three cancellous screws with an inverted triangle pattern are used to fix the fracture of femoral neck.
  Arms: Multiple cancellous screws (MCS)

SUMMARY:
This prospective multicenter cohort study is to compare the post-operative implant failure rate between the patients with femoral neck fracture (AO classification 31-B) using Femoral Neck System (FNS) versus Multiple Cancellous Screws (MCS) at 2-year follow up. The patients are divided into the FNS group and the MCS group according to the internal fixation they choose. The internal fixation failure rate (IFFR) and differences in fracture prognosis of the two groups will be compared. Obtain clinical data of FNS in the Chinese population, and verify the safety and efficacy of FNS for patients with femoral neck fracture.

DETAILED DESCRIPTION:
This is a prospective multicenter cohort study. The team leader is Peking University Third Hospital. All patients are divided into 2 groups according to the internal fixation they choose. Investigators use FNS for internal fixation in Group 1 and MCS in Group 2. Since FNS is clinically comparable to the Dynamic Hip Screw (DHS) system, investigators used DHS clinical data as a statistical reference. The relevant parameters of the sample calculation are α = 0.05 (one-sided) and β = 0.2. PASS 15 was used for calculation, and the final sample size was 290. The FNS group and the MCS group each included 145 patients. See the text for detailed inclusion and exclusion criteria. Patients that meet all the inclusion criteria but do not meet any exclusion criteria, and who have signed the informed consent will be recruited, and each patient will be assigned a unique patient identification number, which will be used throughout the study identify the patient. Investigators will perform preoperative preparation, intraoperative operation and internal fixation implantation according to the instructions provided in the product packaging. Investigators only plan to include cases that can successfully conduct closed reduction, therefore investigators will exclude cases that require open reduction. For the MCS group, three cancellous screws with an inverted triangle pattern are used to fix the fracture of femoral neck. After the operation, the patients will be managed according to the standard nursing and rehabilitation procedures of the experimental site and the results of laboratory tests will be recorded. Regular follow-up evaluation will be performed after the operation until the end of the two-year follow-up or the primary end point of the study. In this study, the internal fixation failure rate (IFFR) is used as the primary end point of the study, which is defined as the total incidence of internal plant cut-out and fracture. The results of the radiographic examination, the lateral X-ray film and computed tomography(CT), will be evaluated by an independent radiologist to determine whether there are cut-out or fracture of the internal plant. Secondary endpoints include: 1. Bone nonunion after 36 weeks: evaluate bone healing according to the lateral X-ray examination. According to the regulations of Food and Drug Administration of the US, it is defined as nonunion if there are no obvious signs of fracture healing 9 months after the fracture, or if there is no obvious difference in fracture space after three consecutive months. 2. Garden classification proportion, and Garden index for reduction assessment. 3. Clinical prognosis: o A 12-Item Short-Form Health Survey (SF-12) o Harris hip score. 4. Operation time, from the incision to internal fixation implanted. 5. The times of intraoperative fluoroscopy, average 25 milliseconds per X-ray shot, record the number of X-ray shot. 6. Postoperative adverse events within 2 years, including ipsilateral femoral head avascular necrosis, infection, wound hematoma, ipsilateral coxa vara, and ipsilateral limb shortening. In this study, it is difficult to blind anyone . Investigators will try their best to reduce human-induced bias in experimental results. Investigators will use one-sided α = 0.05 for statistical tests and confidence interval calculations. P value <0.05 is considered statistically significant. SPSS (latest version: SPSS Inc., Chicago, IL, USA) will be used to analyze the results.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients with unilateral femoral neck fractures that will be treated with internal fixation
3. According to AO fracture classification, subjects with the fracture type (31-B)
4. Subjects (with the help of relatives) can understand the informed documents and patient questionnaires.
5. Subjects (with the help of relatives) voluntarily provide written informed consent to participate in the clinical study and authorize the transfer of their information to the sponsor.
6. The investigator believes that the subject can understand the clinical study, is willing and able to complete all research procedures and follow-up visits and can cooperate with the research procedures.
7. In-label use of the MCS and FNS.

Exclusion Criteria:

1. Subject does not provide voluntary consent to participate in the study.
2. The researcher believes that the subjects have conditions that affect the participation and follow-up of this study. (for example, the patient lives in a remote area or has difficulty in going back to the hospital for follow-up or does not cooperate with the medical guidance and suggestions of the surgeon.)
3. The subjects were pregnant or lactating women.
4. The researchers believe that the subjects have psychological disorders, which may affect the treatment outcome.
5. Garden classification III and IV of femoral neck fracture patients older than 65 years
6. Concurrent hip osteoarthritis.
7. Fractures where the operative treatment will occur more than three weeks after the primary injury
8. Patients combined with other bone fractures.
9. Pathological fracture (e.g., primary or metastatic tumor)
10. Serious soft tissue injury, judged by the investigator, will impact the union of the fracture, combined open fractures, vascular injury, and combined osteofascial compartment syndrome
11. Multiple systemic injuries judged by researchers not suitable for enrollment.
12. Revision surgeries (for example, due to malunion, nonunion or infection)
13. Concurrent medical conditions judged by researchers not suitable for enrollment, such as: metabolic bone disease, post-polio syndrome, poor bone quality, prior history of poor fracture healing, etc
14. Patients with anaesthetic and surgical contraindications
15. Patients known to be allergic to implant components
16. Patients who are currently using chemotherapeutics or accepting radiotherapy, use systematically corticosteroid hormone or growth factor, or long-term use sedative hypnotics (continuous use over 3 months) or non-steroidal anti-inflammatory drugs (continuous use over 3 months)
17. Intemperance judged by researchers not suitable for enrollment (e.g., excessive daily drinking or smoking, drug abuse);
18. Subjects participated in other clinical studies in the past 3 months, which may affect the outcome and follow-up according to the judgment of researchers.
19. Subjects have significant neurological or musculoskeletal disorders or may have adverse effects on gait or weight-bearing (e.g., muscular dystrophy, multiple sclerosis, cerebral infarction, hemiplegia, Charcot arthropathy, avascular necrosis of the femoral head).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Internal fixation failure rate | from operation to 2-year follow-up after the surgery
  defined as the total incidence of internal plant cut-out and fracture.

SECONDARY OUTCOMES:
Number of Participants with Bone nonunion | from operation to 2-year follow-up after the surgery
  evaluate bone healing according to the lateral X-ray examination. According to the regulations of Food and Drug Administration of the US, if there are no obvious signs of fracture healing 9 months after the fracture, or if there is no obvious difference in fracture space after three consecutive months, it is defined as nonunion.
Harris hip score | from operation to 2-year follow-up after the surgery
  the score value is from 0 to 100, and a higher score means a better outcome
operation time | intraoperative
  from the incision to internal fixation implanted.
The times of intraoperative fluoroscopy | intraoperative
  average 25 milliseconds per X-ray shot, record the number of X-ray shot
Number of Participants with Postoperative adverse events | from operation to 2-year follow-up after the surgery
  including ipsilateral femoral head avascular necrosis, infection, wound hematoma, ipsilateral coxa vara, and ipsilateral limb shortening
Garden index | from operation to 2-year follow-up after the surgery
  The fracture reduction will be considered unsatisfied if the index is less than 155 degrees or more than 180 degrees.
A 12-Item Short-Form Health Survey (SF-12) | from operation to 2-year follow-up after the surgery
  the score value is from 0 to 100, and a higher score means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Fang Zhou, MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No